CLINICAL TRIAL: NCT03752333
Title: A Phase II, Two-Stage, Trial of Pembrolizumab in Cancer of Unknown Primary
Brief Title: Trial of Pembrolizumab in Cancer of Unknown Primary
Acronym: CUPem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/37/2017
Record Dates: First submitted 2018-11-15; First posted 2018-11-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): All trial treatments will be administered on an outpatient basis. Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab has high affinity and potent receptor blocking activity for PD-1, based on preclinical in vitro data. Pembrolizumab has an acceptable preclinical and clinical safety profile and is in clinical development as an IV immunotherapy for advanced malignancies.
  The PD-1 pathway represents a major immune control switch, which may be engaged by tumour cells to overcome active T-cell immune surveillance. Pembrolizumab is a potent and highly selective humanized mAb of the Immunoglobulin (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. This blockade enhances functional activity of the target lymphocytes to facilitate tumor regression and ultimately immune rejection.
  Other Names: Keytruda

SUMMARY:
Abbreviated Title : CUPem Clinical Indication : A Phase II, Two-Stage, Trial of Pembrolizumab in Cancer of unknown primary Trial Type : Single Arm, non-randomised; Two-stage; Hypothesis generating Type of control : None Route of administration : IV Trial Blinding : N/A

Treatment Groups :Two cohorts:

(i) First Cohort: One or more lines of prior therapy (ii) Second Cohort: First Line untreated CUP patients Number of trial subjects : i) First Cohort: 20 ii) Second Cohort: 57 Eligibility Criteria : The Eligibility Criteria are the same as used in the A trial of chemotherapy for cancer of unknown primary (CUP-ONE) trial in the United Kingdom (UK), please see below.

* Histologically confirmation of a diagnosis of CUP, with imaging and all diagnostic investigations confirmed as CUP within a CUP Multidisciplinary Team (MDT).
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Patients must have disease that is not amenable to potentially curative options such as resection or radical radiotherapy
* If patient's disease presentation precludes tumour biopsy (inaccessible or biopsy thought not to be in the patient's best interest), the patient is not study eligible.

Estimated recruitment period : 2 years Estimated duration of trial : 3.9 years including set up, recruitment, follow up and close down.

Duration of Participation : Cohort 1 = 6-8 months; Cohort 2 = 8-18 months Estimated average length of treatment per patient =6 months

DETAILED DESCRIPTION:
An open label, non-randomised, single arm, sequential phase (two sequential cohorts) study, evaluating the preliminary efficacy of Pembrolizumab in Cancer of unknown Primary (CUP).

Cohort 1:

Cohort 1 will enrol a maximum of 20 patients, who have had at least one prior line / regimen of chemotherapy (at least 2 cycles) appropriate for CUP and who have not had a RECIST response to first-line chemotherapy, or are progressing after an initial response, or are treatment intolerant to first-line chemotherapy, due to unacceptable toxicity.

As soon as there has been one documented response in cohort 1, the study then proceeds to enrol cohort 2 in parallel. Cohort 2 will not be initiated, if have been no cohort 1 (0/20) patients who have benefitted and 20 cohort 1 patients have completed at least 12 weeks of therapy. Benefit for this study is defined as either a RECIST or irRECIST response; stable disease for a minimum of 12 weeks. This allows a go / no-go decision to proceed/ not proceed to enrolling cohort 2 by the trial management group

Cohort 2:

Cohort 2 will enrol a maximum of 57 patients who are chemo-naïve (first-line setting) for CUP*, with a PS 0-2. Benefit for this study is defined as either a RECIST or irRECIST response or stable disease at 12 weeks.

*Previous chemotherapy for other cancers is allowed

For both cohorts, patients will undergo screening procedures during a standard 28-days time window from initiation of the study, under standard Good Clinical Practice (GCP) and informed consent. Restaging will be performed by computerized tomography using ir-RECIST criteria at 3 months from initiation of systemic treatment and on an 8 weekly basis thereafter until radiological proven disease progression or intolerance or patient choice.

The EORTC Quality of Life Questionnaire (QLQ-C30) questionnaire (to assess the quality of life) will be done at baseline after 3 months and then at discontinuation of study treatment.

Correlative translational study samples (blood) and tissue (used for histological confirmation and to document Programmed Death-Ligand 1 (PD-L1) expression) will be collected at baseline, and blood and serum samples monthly (after an informed optional consent and banked for retrospective immune-modulating and other biomarkers for future research and analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1
4. Be willing to provide consent for archival tumour (in the form of formalin fixed paraffin embedded (FFPE) block) or fresh tumour material (if judged technically feasible by radiologist is mandatory for diagnosis and biomarker analysis.
5. Have a performance status of 0-2 on the ECOG Performance Scale.
6. Cohort 1 - have had at least one prior line / regimen of chemotherapy appropriate for CUP (at least 2 cycles), have not had a RECIST response to first-line chemotherapy, or are progressing after an initial response, or are treatment intolerant to first-line chemotherapy, due to unacceptable toxicity.

   Cohort 2 - be chemo-naive for CUP*

   *Previous chemotherapy for other cancers is allowed
7. Adequate organ and bone marrow function (all screening tests should be performed within 10 days of treatment initiation):

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Haemoglobin ≥ 9 g/dL (≥90 g/L) without transfusion or Erythropoietin (EPO) dependency (within 7 days of assessment)
   4. Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN) or Creatinine clearance* ≥ 60 mL/min for patients with creatinine levels > 1.5 x ULN

      * Creatinine clearance should be calculated per institutional standard
   5. Serum total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 ULN
   6. Aspartate aminotransferase [AST] ≤ 2.5 x ULN (< 5 x ULN if liver metastases are present)
   7. Alanine aminotransferase [ALT]) ≤ 2.5 x ULN (< 5 x ULN if liver metastases are present)
   8. Albumin ≥ 2.5g/dL
   9. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
   10. Activated Partial Thromboplastin Time (APTT) ≤1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
8. Female subject of childbearing potential should have a mandatory negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 6.9.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 6.9.2 - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis-C Virus (HCV) RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Overall response rates by immune-related (irRECIST) and RECIST criteria in a second-line & first-line setting | 6 months (based on average length of treatment per patient)
  Pembrolizumab has Efficacy in CUP
  * as a first-line treatment in terms of Response which translates into improved progression-free survival (PFS) and overall survival (OS)
  * as a second-line treatment in terms Response which translates into improved PFS and OS
  * and treatment leads to rapid improvement in QOL in high metastatic disease burden (in any line of therapy)

SECONDARY OUTCOMES:
Incidence of adverse events up to 8 weeks after the last dose of Pembrolizumab in the second line setting | 6-8 months (based on average length of treatment per patient
  Pembrolizumab is much better tolerated than conventional chemotherapy in CUP patients and PS2 patients may also benefit.
Incidence of adverse events up to 8 weeks after the last dose of Pembrolizumab in Performance Status 2 (PS2) patients in any setting | 6-8 months (based on average length of treatment per patient)
  • Pembrolizumab is much better tolerated than conventional chemotherapy in CUP patients and PS2 patients may also benefit.

OTHER OUTCOMES:
Identification of potential genomic biomarkers predictive of immune response to Pembrolizumab | 12 months (post study completion)
  This would be a retrospective analysis of blood samples collected for future research purposes only. Research bloods will be used to examine DNA and measure various blood biomarkers. These biomarkers may predict possible response to study treatment. As these samples are being taken before, during and after treatment, they will help us understand how the study treatments work. This will also enable us to learn whether or not the treatments have the desired effect, and to understand if these effects may be beneficial for the treatment of cancer of unknown primary (CUP). This information may also be used to develop and test other new treatments in the future. The panel of potential biomarkers against which the blood plasma will be tested has not been established yet. Information gained from this research component is not directly beneficial to patients taking part in this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet Wasan, MBBS, FRCP, Study Chair — Imperial College London
Locations (3):
- United Kingdom (3):
  - Gastrointestinal Units - The Royal Marsden Hospitals at Sutton and London, Sutton, Surrey
  - Hammersmith Hospital, London
  - Guy's Cancer Centre, London

IPD SHARING:
Plan to Share IPD: Undecided